CLINICAL TRIAL: NCT02502864
Title: Multicenter Study Investigating Utilization of Pharmacokinetic(PK)-Guided Docetaxel in Senior Adult Breast Cancer Patients Receiving Docetaxel and Cyclophosphamide (TC) Chemotherapy
Brief Title: Multicenter Study of Pharmacokinetic-Guided Docetaxel in Breast Cancer Patients Receiving Docetaxel and Cyclophosphamide
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Saladax Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-18118
Record Dates: First submitted 2015-07-15; First posted 2015-07-20 (Estimated); Results first posted 2018-10-18 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Breast Cancer; Breast Cancer Female
Keywords: senior adult; postmenopausal
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Cyclophosphamide; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Standard of Care + Surveys (Experimental): Standard of Care Docetaxel and Cyclophosphamide (TC) Chemotherapy + Surveys. TC Regimen with Function Assessment of Cancer Therapy (FACT) Surveys. All participants will receive TC for cycle 1 with subsequent cycles repeated every 3 weeks for a total of 4 cycles. All initial dosing will be based on actual body weight and height. Participants will receive up to 4 doses of chemotherapy. Following their 4th dose of chemotherapy, or the last dose of chemotherapy in which blood level monitoring was performed, participants will be assessed for side effects from the chemotherapy and complete their final written 53 question survey about their quality of life.
  Interventions: Drug: Standard of Care: Docetaxel; Drug: Standard of Care: Cyclophosphamide; Other: Function Assessment of Cancer Therapy (FACT) Surveys

INTERVENTIONS:
Drug: Standard of Care: Docetaxel — Pharmacokinetic(PK)-guided docetaxel. Cycle 1: 75 mg/m^2, intravenously (IV) on Day 1 for 60 minutes. Beginning with cycle 2, the docetaxel dose will be individually adjusted before each cycle.
  Other Names: Taxotere®
Drug: Standard of Care: Cyclophosphamide — Cycle 1: 600 mg/m^2, via IV on Day 1 for 30 minutes. The cyclophosphamide dose will not be changed unless dictated by toxicity.
  Other Names: Cytoxan®
Other: Function Assessment of Cancer Therapy (FACT) Surveys — Participants will complete the FACT-Taxane and FACT-Breast quality of life assessment written surveys at baseline, during each chemotherapy cycle, and 3-5 weeks following the last cycle in which PK monitoring was performed.
  Other Names: Questionnaire

SUMMARY:
The purpose of this study is to adjust the amount of docetaxel participants receive based on the level of docetaxel measured in their blood. This method of dose adjustment is called pharmacokinetic (PK)-adjusted docetaxel. The researchers believe that adjusting the dose of docetaxel using this method will lessen the side effects associated with docetaxel in cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Must have histologically confirmed localized or locally advanced breast cancer for which the treatment plan includes chemotherapy with 4 cycles of standard TC (docetaxel 75 mg/m^2 and cyclophosphamide 600mg/m^2)
* Age >/= 65 years (Senior adult focused study given increased risk for toxicity)
* Participants must be female
* Eastern Cooperative Oncology Group (ECOG) performance status <2
* Must have normal organ and marrow function
* No pre-existing neuropathy grade > 1 per the NCI Common Toxicity Criteria for Adverse Effects (CTCAE) version 4.0
* Be postmenopausal (defined as amenorrheic for at least 12 months)
* Must be informed of the investigational nature of this study and be willing to provide written informed consent in accordance with Institutional guidelines and Good Clinical Practice (GCP) indicating that they understand the purpose of and procedures required for the study and are willing to participate prior to the beginning of any specific study procedures.

Exclusion Criteria:

* Have uncontrolled illness (including, but not limited to, ongoing or active infection, congestive heart failure, angina pectoris, or cardiac arrhythmia) that would limit compliance with study requirements
* Have psychiatric illness that would limit compliance with study requirements
* Have history of allergic reactions attributed to compounds of similar chemical or biologic composition to taxanes (docetaxel or paclitaxel) or cyclophosphamide
* Have known seropositivity for human immunodeficiency virus, hepatitis C virus, hepatitis B surface antigen, or syphilis. Does not require serologic confirmation as a study procedure.
* Not willing to follow protocol requirements or to give informed consent

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-02-09 (Actual); Primary Completion 2017-09-29 (Actual); Study Completion 2019-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Walko, Pharm.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at Moffitt Cancer Center, February 2016 through June 2017.
Period: Overall Study
Arm/Group | Standard of Care + Surveys
Started | 9
Completed | 8
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: All participants.
Groups:
- Standard of Care + Surveys: Standard of Care Docetaxel and Cyclophosphamide (TC) Chemotherapy + Surveys. TC Regimen with Function Assessment of Cancer Therapy (FACT) Surveys.
Arm/Group | Standard of Care + Surveys
Number analyzed (Participants) | 9
Age, Continuous [Mean (Full Range); unit: years] | 72 [66 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Rate of Achieving Targeted Area Under the Curve (AUC)
Description: Rate of PK guided dosing of docetaxel chemotherapy improving the ability to achieve a targeted AUC ( 2.5-3.7 mg*hr/L) within 4 cycles of therapy in patients > 65 years of age with breast cancer receiving TC (docetaxel and cyclophosphamide) as compared with historical non-PK guided therapy from patients receiving a similar regimen.
Time Frame: Cycle 4 - Up to 6 months
Population: All participants evaluable at time of analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care + Surveys
Number analyzed (Participants) | 8
Participants
  AUC mg*hr/L: 2.5-3.7 | 5
  AUC mg*hr/L: <2.5 | 3

2. Secondary Outcome: Incidence of Grade 3 and 4 Neutropenia and Febrile Neutropenia
Description: The incidence of grade 3 and 4 neutropenia and febrile neutropenia in cycles following PK adjustment (cycles 2-4) will be compared with cycle 1 and historical non-PK guided therapy using the Wilcoxon-Rank sum assessment.
Time Frame: Up to 6 months
Population: All participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care + Surveys
Number analyzed (Participants) | 9
Participants
  Participants with Grade 3 or 4 neutropenia | 2
  Participants with Febrile neutropenia | 0

3. Secondary Outcome: Association Between Scores - Chemotherapy Risk Assessment Scale for High-Age Patients
Description: The Chemotherapy Risk Assessment Scale for High-Age Patients (CRASH) score will be reported as ordinal data (low, intermediate-low, intermediate-high, or high risk).
Time Frame: Baseline and Post Cycle 1
Population: Descriptive analysis was planned for 52 participants. Due to the small number of participants enrolled, analyzing additional correlations was not possible.
Arm/Group | Standard of Care + Surveys
Number analyzed (Participants) | 0

4. Secondary Outcome: Association Between Scores - Instrumental Activities of Daily Living
Description: The Instrumental Activities of Daily Living (IADL) total score will be reported as binomial data (greater or less than 26 based on how it is incorporated into the CRASH score).
Time Frame: Baseline and Post Cycle 1
Population: as for outcome 3
Arm/Group | Standard of Care + Surveys
Number analyzed (Participants) | 0

5. Secondary Outcome: Association Between Scores - Cumulative Illness Rating Scale for Geriatrics
Description: The Cumulative Illness Rating Scale for Geriatrics (CIRS-G) will be reported as discrete data out of a possible score of 65. The Wilcoxon-Rank sum and Chi-squared tests will be used as appropriate.
Time Frame: Baseline and Post Cycle 1
Population: as for outcome 3
Arm/Group | Standard of Care + Surveys
Number analyzed (Participants) | 0

6. Other Pre Specified Outcome: Comparison of Patient Profiles and Function Assessment of Cancer Therapy (FACT) Scores
Description: The relationship between PK-guided docetaxel patient PK profiles and the Function Assessment of Cancer Therapy (FACT) Taxane and Breast Cancer scores will be described.
Time Frame: Up to 6 months
Population: as for outcome 3
Arm/Group | Standard of Care + Surveys
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year, 9 months
Arm/Group | Standard of Care + Surveys
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 3/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care + Surveys (N=9)
Fatigue (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care + Surveys (N=9)
Constipation (Gastrointestinal disorders) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 5 (8)
Nausea (Gastrointestinal disorders) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Salivary duct inflammation (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 9 (15)
Edema limbs (General disorders) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 6 (7)
Bone pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 4 (6)
White blood cell decreased (Investigations) | 4 (4)
Alkaline phosphatase increased (Investigations) | 2 (2)
Lymphocyte count decreased (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 2 (2)
Creatinine increased (Investigations) | 1 (2)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 3 (3)
Hypertension (Vascular disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Watering eyes (Eye disorders) | 1 (1)
Papulopustular rash (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (2)
Anxiety (Psychiatric disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Recruiting ended early due to slow enrollment. Larger studies may help elucidate a more optimal AUC range for senior adults receiving docetaxel as part of the TC regimen for breast cancer to balance both toxicity and efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-02): https://cdn.clinicaltrials.gov/large-docs/64/NCT02502864/Prot_SAP_000.pdf